CLINICAL TRIAL: NCT01573728
Title: Role of Exercise in Depression Among Middle Aged and Older Adults
Brief Title: Role of Exercise in Depression in Middle Aged and Older Adults
Acronym: RED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Daniel Clark, Associate Professor of Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1111007450; R24MH080827 (NIH)
Record Dates: First submitted 2012-04-05; First posted 2012-04-09 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Depression
Keywords: Depression; Biomarkers; Exercise
MeSH Terms: conditions — Depression; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low Exercise Arm (Active Comparator): Low dose exercise (50 Minutes)
  Interventions: Behavioral: Low dose exercise
- Public Health Exercise (Experimental): Public Health dose exercise (150 minutes)
  Interventions: Behavioral: Public Health Exercise

INTERVENTIONS:
Behavioral: Low dose exercise — Exercise totaling 50 minutes per week and low intensity
  Arms: Low Exercise Arm
Behavioral: Public Health Exercise — At least 150 minutes at moderate intensity
  Arms: Public Health Exercise

SUMMARY:
The pilot project proposed here will establish the feasibility and preliminary data necessary to test in a subsequent randomized trial: 1) whether independent of social contact, aerobic exercise training is effective in the treatment of depression and 2) whether changes in biological markers indicate an anti-inflammatory process, neurogenesis process, or both as a result of exercise. Target participants are adults aged 46 years or over who have current minor to moderate depressive symptoms.

This pilot is a three-arm design of low dose exercise versus public health dose exercise intended to: 1) establish the feasibility, acceptance, and safety of Internet-based supervised exercise training and 2) obtain retention and attendance estimates needed to determine sample sizes for the follow-up trial.

DETAILED DESCRIPTION:
Recruitment will occur by phone or in the clinic by the Practice Based Research Network (PBRN) using the attached screener. Prior to contact, patients will have been identified as potentially eligible by having had a current or past diagnosis of depression as indicated in the Regenstrief Medical Records System. These potentially eligible persons must then be approved for the study and moderate-intensity exercise by their primary care provider before the recruitment call and screener from the PBRN. The telephone screener uses the PHQ 9 (Patient Health Questionnaire-9) and a modified Stanford Brief Physical Activity Scale. Those with a PHQ-9 score of 10 or greater and who indicate no current regular physical activity will be eligible for further screening.

Following recruitment by the PBRN, study personnel will call and confirm the PHQ-9 results with the SCID. If the patient passes the follow-up screening, the staff will arrange to travel to the patient's home. Study staff will obtain informed consent and perform baseline assessments including the Short Form-36, PHQ-9, Generalized Anxiety Disorder-7 (GAD-7), Medical Outcomes Study Social Support survey, and the ASA 24. The ASA 24 is an online dietary screener that measures energy intake over a 24 hour period. It is posted on the National Cancer Institute's website. Medication adherence and smoking levels will be measured by self report. Height, weight, waist circumference, and blood pressure will also be measured. With the exception of the SCID, each of these measures will be repeated at 3 month follow-up. The PHQ-9 will be completed monthly. Also, each month (three different time periods) participants will be asked to wear an armband accelerometer to measure energy expenditure over a 2 week period. The protocol gives details of the accelerometry procedures.

Blood will be drawn using a 2 ten ml tubes at base line and 3 month follow-up using procedures described in the Data Safety and Monitoring Plan. We will ask that the participants fast for eight hours prior to the blood draw, but will note if that was not possible. Appointments for the blood draw will be made within five days of the assessment and also take place within the participant's home.. The blood samples will measure circulating levels of the proinflammatory cytokines IL-1α, IL-1β, IL-6, and TNF-α; the anti-inflammatory cytokines IL-1ra and IL-10; the acute-phase reactant CRP; and VEGF and BDNF.

Participants will be randomized to public health or low dose exercise. Randomization will be stratified by baseline use/no use of prescription anti-depressants. Both low and public health exercise arms will receive supervised one on one instruction via video conference. The exercise will occur five times a week for 10 to 30 minutes each session. During the twelve week intervention, the exercise will increase in intensity and may include wrist and ankle weights. During each session, the participant will rate their perceived exertion using the Borg's Rating of Perceived Physical Exertion (RPE): a 10 Point Scale where 0 is no movement and 10 is maximum effort. Participants will also wear a heart rate monitor. Participants in the low dose exercise arm will be instructed to exercise at an RPE of less than 5 and a heart rate of less than 50% of their age-adjusted maximum (200 minus participant's age). The participants in the public health dose arm will be instructed to exercise at an RPE of between 5 and 7 and to maintain a heart rate of 55 to 70% of age-adjusted maximum heart rate.

All assessments and blood draws will occur in the participant's home.

ELIGIBILITY:
Inclusion Criteria:

46 or older English speaking Community dwelling Access to a private room Access to a telephone Permanent address Willingness to be randomized Internet-enabled computer in home or willingness to have such installed Score of 10 or more on PHQ-9 Major depressive disorder as indicated by the Structured Clinical Interview for DSM-IV (SCID) Primary care provider approval for participation in moderate-intensity exercise

Exclusion Criteria:

Any serious medical condition for which exercise is contraindicated by the ACSM Current diagnosis of one of the following: psychosis, bipolar disorder, lupus, HIV, AIDS, IBS, Crones, Rheumatoid Arthritis or related conditions, cancer or treatment for cancer within the last year. Acute illness Terminal illness (not expected to live beyond one year) Unwillingness to provide informed consent Unwillingness to donate blood Receiving disability insurance Currently engaged in professional psychotherapy Currently engaged in regular exercise Pregnant or nursing in the past 6 months, or plans to become so within 12 months Enrolled in another study Member of household enrolled in the same study Residence outside of Marion County Residence relocation plans within 12 months Substance abuse Suicide ideation as indicated by the PHQ-9

Min Age: 46 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-05; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
PHQ 9 depression score | 3 months

SECONDARY OUTCOMES:
Biomarkers of inflammation and neurogenesis | 3 months
SF-36 | 3 months
Blood Pressure | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel O Clark, PhD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States